CLINICAL TRIAL: NCT07211802
Title: Utilizing Continuous Ketone Monitors to Enable Safe Use of SGLT Inhibitors in Patients With Type 1 Diabetes
Brief Title: CKM For Safe Use of SGLT2i in Type 1 Diabetes
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Abbott (Industry); Lexicon Pharmaceuticals (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Jeremy Pettus, MD, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 812125; 1R01DK143381 (Other Grant/Funding Number: NIH); 1U01DK143381 (NIH)
Record Dates: First submitted 2025-06-16; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: Sotagliflozin; SGLT2; Continuous Ketone Monitor; DGK; CKM
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment Group A (Experimental): 200mg sotagliflozin for 6 weeks, washout for 2 weeks, then receive 400mg sotagliflozin for 6 weeks
  Interventions: Drug: Sotagliflozin Low Dose; Drug: Sotagliflozin High Dose; Device: Dual Continuous Glucose and Ketone Monitor
- Treatment Group B (Experimental): 400mg sotagliflozin for 6 weeks, washout for 2 weeks, then receive 200mg sotagliflozin for 6 weeks
  Interventions: Drug: Sotagliflozin Low Dose; Drug: Sotagliflozin High Dose; Device: Dual Continuous Glucose and Ketone Monitor

INTERVENTIONS:
Drug: Sotagliflozin Low Dose — 200 mg Sotagliflozin, once daily for 6 weeks
Drug: Sotagliflozin High Dose — 400 mg Sotagliflozin, once daily for 6 weeks
Device: Dual Continuous Glucose and Ketone Monitor — Abbott Libre X dual continuous glucose and ketone monitor (DGK) device.

SUMMARY:
This research study is being conducted to learn if wearing a combination continuous glucose monitor/continuous ketone monitor (CGM/CKM) can reduce the side effects of taking sotagliflozin (study drug) in people with type 1 diabetes.

DETAILED DESCRIPTION:
The study is a phase 3, single-site, double-blind, random-order, cross-over study to evaluate the use of continuous ketone monitoring (CKM) in participants with type 1 diabetes taking sotagliflozin.

There will be 2 main groups in the study, participants on Hybrid Closed Loop insulin pumps (HCL), n=26, and participants on Multiple Daily Injections (MDI), n=26. There will also be 2 doses of sotagliflozin examined in the study, 200 milligram (mg) once daily and 400mg once daily. Therefore, there will be 4 treatment groups in the study:

* MDI participants who receive 200mg sotagliflozin for 6 weeks, washout for 2 weeks, then receive 400mg sotagliflozin for 6 weeks;
* MDI participants who receive 400mg sotagliflozin for 6 weeks, washout for 2 weeks, then receive 200mg sotagliflozin for 6 weeks;
* HCL participants who receive 200mg sotagliflozin for 6 weeks, washout for 2 weeks, then receive 400mg sotagliflozin for 6 weeks;
* HCL participants who receive 400mg sotagliflozin for 6 weeks, washout for 2 weeks, then receive 200mg sotagliflozin for 6 weeks.

In addition, there will be an open-label extension study for the HCL group. In the extension study, the 26 participants in the HCL group will remain on their insulin pump, receive a low-dose, open-label, once daily injection of long-acting insulin and complete an additional 6 weeks of dosing with open-label 400 mg sotagliflozin.

For MDI participants there will be a total of 12 visits over approximately 22 weeks. For HCL participants there will be a total of 16 visits over approximately 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. All individuals between the ages of >18 years old, inclusive, at the time of screening;
2. Individuals able to become pregnant must:

   1. be ≥1 year post-menopausal or documented as being surgically sterile, or
   2. agree to use two methods of contraception during the entire study and for an additional 2 weeks after the end of dosing with the investigational product;
3. Individuals able to cause a pregnancy must be willing to use clinically acceptable method of contraception during the entire study and for an additional 2 weeks after the end of the treatment period;
4. Diagnosed with Type 1 diabetes ≥ 1 year prior to screening, based on clinical history or as defined by the current American Diabetes Association (ADA) criteria;
5. Treatment with a stable insulin regimen for at least 8 weeks before screening with:

   1. a continuous subcutaneous insulin infusion (CSII) via a hybrid closed loop system, or
   2. multiple daily insulin injections;
6. Currently using a Continuous Glucose Monitoring (CGM) system;
7. Hemoglobin A1c ≤10% at the time of screening;
8. Estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2;
9. Agrees and is able to wear the investigational device;
10. Able to provide written informed consent approved by an Institutional Review Board (IRB).

Exclusion Criteria:

1. Individuals who are currently pregnant or lactating/breastfeeding, or planning to become pregnant within 10 months after screening;
2. Any concurrent diagnosis of diabetes other than type 1 diabetes;
3. History or evidence of clinically significant disorder or condition that, in the opinion of the Investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures, or completion;
4. Hypotension at screening as defined as, systolic blood pressure < 90 and diastolic blood pressure < 60 with symptoms of low blood pressure (confusion, dizziness, lightheadedness, fainting, heart palpitations);
5. Current or recent (within 1 month prior to screening) use of diabetes medications other than insulin; (examples include, Sodium-Glucose Cotransporter 2 (SGLT-2i), Pramlintide, Metformin);
6. Use of glucagon-like-peptide 1 (GLP-1) analogues if not on a stable dose for > 2 months at screening (participants can be rescreened after being on stable dose for > 2 months). Participants on a stable dose of GLP-1 receptor antagonist (RA) and not experiencing frequent vomiting may be included.
7. Chronic systemic corticosteroids use ( > 4 consecutive weeks) within 6 months prior to screening;
8. History of diabetic ketoacidosis within 3 months prior screening;
9. History of a level 3 hypoglycemic event (as defined by ADA criteria) within 3 months of screening.

   * ADA Level 3 Definition - A severe hypoglycemic event characterized by altered mental or physical status requiring the assistance for treatment of hypoglycemia, irrespective of glucose level;
10. History of multiple (≥3 infections) genital mycotic infections within 6 months of screening;
11. Unable or unwilling to follow the study protocol or who are non-compliant with screening appointments or study visits;
12. Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
BHB Time Above 0.6mmol/L - 200mg | 6 weeks
  Beta hydroxybutyrate (BHB) time > 0.6 millimole per liter (mmol/L) as measured by the DGK during the 200mg dosing period in the MDI vs. HCL groups.
BHB Time Above 0.6mmol/L - 400mg | 6 weeks
  Beta hydroxybutyrate (BHB) time > 0.6 mmol/L as measured by the DGK during the 400mg dosing period in the MDI vs. HCL groups.

SECONDARY OUTCOMES:
BHB Time Above 0.6mmol/L - 200mg vs. 400mg | 6 weeks
  Beta hydroxybutyrate (BHB) time > 0.6 mmol/L as measured by the DGK comparing the 200mg treatment period to the 400mg treatment period.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD - Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No